CLINICAL TRIAL: NCT00064116
Title: Randomized Intergroup Trial of First Line Treatment for Patients With Diffuse Large B-Cell Non-Hodgkin's Lymphoma With a CHOP-Like Chemotherapy Regimen With or Without the Anti-CD20 Antibody Rituximab
Brief Title: Combination Chemotherapy With or Without Rituximab in Non-Hodgkin's Lymphoma
Acronym: IDEC-C2B8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY9; CAN-NCIC-LY9; ROCHE-CAN-NCIC-LY9 (Other: Roche); MINT-M39045; CDR0000309053 (Other: PDQ)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; VAP-cyclo protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: CHOP-21 (Active Comparator): Cyclophosphamide 750 mg/m² i.v. day 1 Doxorubicin 50 mg/m² i.v. day 1 Vincristine 2 mg (abs.) i.v. day 1 Prednisone 100 mg/d p.o. days 1 to 5 Recycle: day 22 Total number of cycles 6
  Interventions: Drug: CHOP regimen
- Arm B: CHOP-21 + Rituximab (Active Comparator): Rituximab 375 mg/m² i.v. day 1* Cyclophosphamide 750 mg/m² i.v. day 1 Doxorubicin 50 mg/m² i.v. day 1 Vincristine 2 mg (abs.) i.v. day 1 Prednisone 100 mg/d p.o. days 1 to 5 Recycle day 22 Total number of cycles: 6
  Interventions: Biological: rituximab; Drug: CHOP regimen

INTERVENTIONS:
Biological: rituximab — Rituximab 375 mg/m² i.v. day 1
  Arms: Arm B: CHOP-21 + Rituximab
Drug: CHOP regimen — Cyclophosphamide 750 mg/m² i.v. day 1 Doxorubicin 50 mg/m² i.v. day 1 Vincristine 2 mg (abs.) i.v. day 1 Prednisone 100 mg/d p.o. days 1 to 5 Recycle day 22 Total number of cycles: 6

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy is more effective with or without rituximab in treating patients with non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying four different combination chemotherapy regimens and rituximab to see how well they work compared to four different combination chemotherapy regimens alone in treating patients with non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to treatment failure in patients with CD20-positive diffuse large B-cell non-Hodgkin's lymphoma treated with CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisone)-like chemotherapy with vs without rituximab.
* Compare the tumor control, progression rate, and complete remission rate in patients treated with these regimens.
* Compare the disease-free and overall survival rate of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center, bulky disease (no vs yes), International Prognostic Index score (0 vs 1), and chemotherapy (CHOP vs CHOEP vs PMitCEBO vs MACOP-B). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive 1 of the following chemotherapy regimens according to participating country:

  * CHOP: Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisone or prednisolone on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  * CHOEP-21: Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1; etoposide IV on days 1-3; and oral prednisone on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  * PMitCEBO: Patients receive mitoxantrone IV, cyclophosphamide IV, and etoposide IV on day 1; vincristine IV and bleomycin IV on day 8; and oral prednisolone daily during weeks 1-4 and every other day during week 5. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  * MACOP-B: Patients receive cyclophosphamide IV and doxorubicin IV on days 1, 15, 29, 43, 57, and 71; methotrexate IV and vincristine IV on days 8, 36, and 64; bleomycin IV and vincristine IV on days 22, 50, and 78; and oral or intramuscular prednisone on days 1-84. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive arm I regimens (according to participating country) and rituximab as follows:

  * CHOP and rituximab: Patients receive CHOP as in arm I and rituximab IV on day 1.
  * CHOEP-21 and rituximab: Patients receive CHOEP-21 as in arm I and rituximab IV on day 1.
  * PMitCEBO and rituximab: Patients receive PMitCEBO as in arm I and rituximab IV on day 1 during courses 1 and 4; on day 8 during courses 2 and 5; and on day 1 at 1 and 4 weeks after completion of the last course of PMitCEBO chemotherapy.
  * MACOP-B and rituximab: Patients receive MACOP-B as in arm I and rituximab IV on days 1, 22, 43, 64, 85, and 106.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 820 patients will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell non-Hodgkin's lymphoma according to REAL classification

  * Diagnosed within the past 6 weeks
  * CD20+ disease
  * Ann Arbor stage II, III, or IV disease or stage I bulky disease
* International Prognostic Index (IPI) score of 0 or 1

  * Score 0 defined by all of the following:

    * Stage I or II disease
    * ECOG performance status of 0 or 1
    * Lactic dehydrogenase (LDH) no greater than upper limit of normal (ULN)
  * Score 1 defined by 1 of the following:

    * Stage I or II disease; ECOG performance status of 0 or 1; and LDH greater than ULN
    * Stage I or II disease; ECOG performance status 2 or 3; and LDH no greater than ULN
    * Stage III or IV disease; ECOG performance status 0 or 1; and LDH no greater than ULN
* Previously untreated disease
* Mediastinal B-cell lymphoma allowed
* No secondary lymphoma after prior chemotherapy or radiotherapy for other malignancies
* No transformed lymphoma
* No primary CNS lymphoma
* No primary gastrointestinal (MALT) lymphoma
* No post-transplant lymphoproliferative disorder

PATIENT CHARACTERISTICS:

Age

* 18 to 60

Performance status

* See Disease Characteristics
* ECOG 0-3

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2.0 mg/dL*
* Transaminases no greater than 3 times normal*
* No active chronic hepatitis B or C infection NOTE: *Unless related to lymphoma

Renal

* Creatinine no greater than 2 times normal* NOTE: *Unless related to lymphoma

Cardiovascular

* No myocardial infarction within the past 6 months
* No uncompensated heart failure
* No dilatative cardiomyopathy
* No coronary heart disease with ST segment depression on ECG
* No severe uncompensated hypertension

Pulmonary

* No chronic lung disease with hypoxemia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No known allergic reactions against foreign proteins
* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No concurrent disease that would preclude study treatment
* No active infections requiring systemic antibiotics or antiviral medications
* No severe uncompensated diabetes mellitus
* No clinical signs of cerebral dysfunction
* No severe psychiatric disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior murine antibodies

Chemotherapy

* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent response-adapted (slow response or unconfirmed complete response) radiotherapy

Surgery

* Not specified

Other

* No prior lymphoma-specific treatment
* More than 12 weeks since prior participation in another clinical trial
* No prior participation in this study
* No other concurrent study medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 824 (Actual)
Dates: Start 2001-05-08 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2014-01-16 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) at 3 years | 3 years

SECONDARY OUTCOMES:
Complete remission rate after completion of treatment | 3 years
Overall survival at 3 years | 3 years
Tumor control measured by TTF with non-tumor events censored at 3 years | 3 years
Disease-free survival (DFS) measured by TTF after an event during and directly after treatment at 3 years | 3 years
Progression rate determined by dividing the number of patients with disease progression by number of patients with evaluable outcome at 3 years | 3 years
Time to progression measured at 3 years | 3 years
Toxicity assessed by NCI CTC v2.0 after completion of treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Imrie, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (25):
- Canada (25):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-The Toronto General Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Centre - West Toronto, Toronto, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pfreundschuh M, Ho AD, Cavallin-Stahl E, Wolf M, Pettengell R, Vasova I, Belch A, Walewski J, Zinzani PL, Mingrone W, Kvaloy S, Shpilberg O, Jaeger U, Hansen M, Corrado C, Scheliga A, Loeffler M, Kuhnt E; MabThera International Trial (MInT) Group. Prognostic significance of maximum tumour (bulk) diameter in young patients with good-prognosis diffuse large-B-cell lymphoma treated with CHOP-like chemotherapy with or without rituximab: an exploratory analysis of the MabThera International Trial Group (MInT) study. Lancet Oncol. 2008 May;9(5):435-44. doi: 10.1016/S1470-2045(08)70078-0. Epub 2008 Apr 8. PMID 18400558
- [Result] Pfreundschuh M, Trumper L, Osterborg A, Pettengell R, Trneny M, Imrie K, Ma D, Gill D, Walewski J, Zinzani PL, Stahel R, Kvaloy S, Shpilberg O, Jaeger U, Hansen M, Lehtinen T, Lopez-Guillermo A, Corrado C, Scheliga A, Milpied N, Mendila M, Rashford M, Kuhnt E, Loeffler M; MabThera International Trial Group. CHOP-like chemotherapy plus rituximab versus CHOP-like chemotherapy alone in young patients with good-prognosis diffuse large-B-cell lymphoma: a randomised controlled trial by the MabThera International Trial (MInT) Group. Lancet Oncol. 2006 May;7(5):379-91. doi: 10.1016/S1470-2045(06)70664-7. PMID 16648042